CLINICAL TRIAL: NCT01079624
Title: Effects of GIP and GLP-1 on Gastric Emptying, Appetite and Insulin-glucose Homeostasis
Brief Title: GIP and GLP-1 on Gastric Emptying, Appetite and Insulin-glucose
Acronym: GIP-GLP-gas
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Uppsala University (Other)
Collaborators: Karolinska Institutet (Other); University of Copenhagen (Other)
Responsible Party: Professor Per Hellström, Uppsala University
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: GIP/GLP-gastric empt-APP-hor; K2010-55X -07916-24-3 (Other Grant/Funding Number: Swedish Research Council)
Record Dates: First submitted 2010-03-02; First posted 2010-03-03 (Estimated); Last update posted 2010-03-03 (Estimated); Status verified 2009-07

CONDITIONS: Physiology; Gastroenterology; Endocrinology
Keywords: Incretin hormones; Glucose-insulinotropic peptide; Glucagon-like peptide-1; Gastric emptying; Appetite; Glucose disposal; Gut hormones
MeSH Terms: interventions — Glucagon-Like Peptide 1; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- GIP two doses and GLP-1 one dose (Experimental): Intervention with infusion of GIP or GLP-1 intravenously
  Interventions: Other: Glucose-insulinotropic peptide, Glucagon-like peptide-1
- Saline infusion (Placebo Comparator): Control
  Interventions: Other: Glucose-insulinotropic peptide, Glucagon-like peptide-1

INTERVENTIONS:
Other: Glucose-insulinotropic peptide, Glucagon-like peptide-1 — GIP 2 and 5 pmol/kg min GLP-1 0.7 pmol/kg min
  Other Names: GIP; GLP-1; Saline

SUMMARY:
Academic phase 1 study which investigates the effects of the two incretin hormones glucose-insulinotropic peptide (GIP) and glucagon-like peptide-1 (GLP-1) on gastric emptying, appetite, insulin release and glucose disposal in the body. The hypothesis is that incretin hormones not only stimulate insulin release but also inhibits gastric emptying. This effect can be utilized for further drug development.

DETAILED DESCRIPTION:
Effects of GIP and GLP-1 on gastric emptying, appetite control and insulin release in relation to glucose levels in the bloodstream. Infusions of GIP and GLP-1 are given under simultaneous gastric emptying study and appetite questionnaires and blood sampling for analysis of insulin, glucose, and other gut hormones such as glucagon, ghrelin, and PYY, as well as those administered, GIP and GLP-1.

ELIGIBILITY:
Inclusion Criteria:

* Men and women
* 18-50 years old;
* otherwise healthy and HIV and HCB, HCV negative

Exclusion Criteria:

* Age >50,
* all types of diseases and drug users.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 15 (Actual)
Dates: Start 2006-08; Primary Completion 2008-01 (Actual); Study Completion 2009-11 (Actual)

PRIMARY OUTCOMES:
Gastric emptying rate | 2005-2006

SECONDARY OUTCOMES:
Plasma glucose, insulin release, appetite | 2005-2006

CONTACTS AND LOCATIONS:
Overall Officials: Per M Hellstrom, MD, PhD, Principal Investigator — Karolinska Institutet, Uppsala University
Locations (1):
- Karolinska University Hospital, Stockholm, Stockholm County, Sweden